CLINICAL TRIAL: NCT02905695
Title: Contribution of the Local Infiltration of Chirocaine® in the Management of the Post-partum Perineal Pain After Episiotomy or First-degree Tear
Brief Title: Post-partum Perineal Pain - Chirocaine®
Acronym: EPISIO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010/44
Record Dates: First submitted 2016-09-11; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Post-partum Perineal Pain; Episiotomy; Vaginal Tear
Keywords: Post-partum Perineal pain; Episiotomy; First-degree tear
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Chirocaine
  Interventions: Drug: Chirocaine
- Group B (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Chirocaine
  Arms: Group A
Other: Placebo
  Arms: Group B

SUMMARY:
The aim of this placebo-controlled clinical trial is to assess the effectiveness of the local infiltration of the analgesic Chirocaïne® on perineal pain after episiotomy or first-degree tear. The pain intensity is measured in immediate postpartum period by using a numerical rating scale (NRS) at the following times: H2, H4, H8, H12, H24, H36, H48 during rest, defecation and during activities. The safety of Chirocaïne® and the patient satisfaction are also evaluated at each time.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Patients aged 18-45 years
* Single pregnancy.
* Vaginal normal birth in cephalic presentation or assisted vaginal delivery by vacuum extractor.
* Patients having a mediolateral episiotomy or a first-degree perineal tear, epidural analgesia.
* Patients affiliated to a national insurance scheme
* Patients who have given their written consent

Exclusion Criteria:

* Patient not speaking, reading, writing French.
* Multiple pregnancy.
* Breech delivery or instrumental delivery by forceps or spatula.
* Intact perineum.
* No epidural analgesia.
* Patient who represent contraindication to local anesthetics, severe arterial hypotension.
* Previous tear requiring sutures.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Post-partum perineal pain measured by a numerical rating scale | 8 hours post partum

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Ayoubi, MD, PhD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No